CLINICAL TRIAL: NCT01738672
Title: Inhaled Nitrous Oxide and Labor Analgesia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Ya'aqov Abrams (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Ya'aqov Abrams, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO11090221
Record Dates: First submitted 2012-11-17; First posted 2012-11-30 (Estimated); Results first posted 2017-11-21 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-10

CONDITIONS: Labor Pain
Keywords: Nitrous oxide; labor and delivery; analgesia
MeSH Terms: conditions — Labor Pain; Agnosia | interventions — Entonox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nitrous Oxide (Experimental): Parturients who request labor analgesia will be offered inhaled nitrous oxide for labor analgesia.
  Interventions: Drug: Inhaled nitrous oxide

INTERVENTIONS:
Drug: Inhaled nitrous oxide — Administration of nitrous oxide for labor analgesia
  Other Names: N2O; Nitronox; Entonox

SUMMARY:
Hypothesis: The administration of nitrous oxide for labor analgesia will decrease the labor epidural anesthesia rate by 15%.

Specific Aim: To determine if nitrous oxide can be an effective alternative technique for the provision of labor analgesia at Magee-Womens Hospital.

DETAILED DESCRIPTION:
Inhalational anesthetic agents have been used since the mid 1800s to help alleviate pain associated with labor. James Simpson and John Snow initially utilized ether and chloroform respectively in 1847 and 1853. Stanislav Klikovich followed in his predecessors footsteps and successfully administered nitrous oxide for labor analgesia in 1881. Although many inhalational agents have been considered for labor analgesia since that time, the administration of nitrous oxide has been refined over the last century and remains a common practice for obstetrical anesthesia today. Since that time, nitrous oxide has been found to be an effective labor analgesia for many women, although providing less pain relief compared then a labor epidural, it has been found to be safe for the mother, baby, and health care providers.

Nitrous oxide is currently used by 60% of laboring women in the United Kingdom, 50% of women who deliver in Australia and nearly 50% of all parturients in Canada and Finland. This compares to a recent article which reported that only two United States hospitals routinely offer nitrous oxide for labor analgesia as the majority of laboring women request an epidural. The epidural rate in the Unites States averages nearly 90% compared to only 14-38% in other parts of the world.

Nitrous oxide is an easy to administer non-flammable, odorless inhalational agent that produces both analgesia and anxiolysis. It is believed the mechanism of action of nitrous oxide is through the release of endogenous opioid peptides into the periaqueductal gray area of the midbrain which stimulates descending noradrenergic pathways resulting in analgesia. These pathways modulate pain in the dorsal horn of the spinal cord through alpha-2 adrenoreceptors. Anxiolytic effects are thought to be caused by inhibition of N-methyl-D-aspartate (NMDA) receptors. In a Swedish study involving 1,997 parturients utilizing inhaled nitrous oxide as the sole anesthetic for labor analgesia, 37.6% of participants reported effective pain relief.

Currently, the rate of labor epidural analgesia at Magee Womens Hospital is approximately 90%. There are many advantages to the use of nitrous oxide for labor analgesia compared to an epidural. Complications associated with labor epidural analgesia can include infection, bleeding, headache, and wet-tap. These complications can result in a prolonged hospital stay that is not associated with the use of nitrous oxide for labor analgesia.

One of the biggest advantages of the use of nitrous oxide for labor analgesia is the significantly lower cost to administer compared to an epidural. In a recent article in the Birth journal, it was noted that the use of nitrous oxide is far less expensive and much simpler than epidural analgesia and does not result in complications requiring additional treatments and prolonged hospital stays. The use of nitrous could have major financial benefits for both Medicaid and private insurance companies. In 2004, the largest cost for these insurance entities was the cost to care for pregnant and laboring women which was reported to cost $41 billion. The most significant cost savings would be the reduction in anesthesia services. Currently average cost per patient for anesthesia staff coverage is 728 dollars. Average re-imbursement for a labor epidural placement is 385 dollars. Nitrous oxide does not require anesthesia staff to implement, saving health care dollars. After the initial investment of the nitrous oxide machine, the only additional cost would be the tubing and mask for the patient and the nitrous oxide and oxygen E-cylinders for delivery.

With Nitrous oxide having many qualities that make it an attractive choice for labor analgesia, many anesthesia providers are questioning its limited use in the United States. It is speculated that it may be cultural issue and that women make decisions regarding labor analgesia based on learned experiences of family and friends, many of whom have not heard of or used nitrous oxide to cope with labor pains. Another reason may be that some authors argue that nitrous oxide is an orphan drug with no pizzazz for professional groups or companies to profit from its use as it causes environmental and occupational hazards which limit its use. No definitive opinion exists to answer this question. Finally, some authors suggest its use is limited due to the disadvantages of nitrous oxide, which include the possibility to cause mood alterations, euphoria, impaired mentation, dysphoria, inappropriate behaviors and nausea and vomiting. These side effects are limited through a number of fail-safe mechanisms built into the nitrous oxide machine which includes the delivery of at least 30% oxygen and 3 liters of fresh gas flow. In addition the proper use includes self administration under direct supervision of a trained provider while the nitrous oxide is in use.

ELIGIBILITY:
Inclusion Criteria:

* all women of childbearing age (including children aged 14 years and above)who are pregnant
* parturients who request labor analgesia of family medicine investigators certified in the use of nitrous oxide for labor analgesia at Magee-Women's Hospital
* informed verbal and written consent

Exclusion Criteria:

* coexisting medical conditions that are contraindications to the use of nitrous oxide (i.e. recent eye or ear surgery, history of Meniere's disease, history of vitamin B-12 deficiency)
* history of severe nausea and vomiting
* history of chronic pain
* inability to hold a facemask
* impairment of consciousness or intoxication at time of delivery
* received intravenous opioids within two hours prior to initiation of nitrous oxide
* impaired oxygenation (ex: lung cysts, pneumothorax, pulmonary hypertension, or pulmonary edema) with a room-air pulse oximetry reading less than 95%
* hemodynamic instability
* non-reassuring fetal heart rate tracing
* inability to read, write and understand the English language enough to complete all survey questionnaires and pain assessment scales.

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ya'aqov Abrams, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nitrous Oxide
Started | 16
Completed | 11
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Nitrous Oxide
Number analyzed (Participants) | 16
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [25 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Labor Pain
Description: Participant reported pain score, using a numerical rating scale (NRS) ranging from no pain (0) to severe pain (10).
Time Frame: At baseline, and at 1 hour after initiation of nitrous oxide
Population: Data are included for all participants from which they were collected.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nitrous Oxide
Number analyzed (Participants) | 16
units on a scale
  Baseline | 8.88 (0.97)
  1 hour after initiation of nitrous oxide: number analyzed (Participants) | 11
  1 hour after initiation of nitrous oxide | 8.18 (1.72)
Statistical Analysis 1: Comparison: Nitrous Oxide; Test type: Other; p = 0.16, t-test, 2 sided

2. Other Pre Specified Outcome: Anxiety
Description: Participant reported anxiety score, using a numerical rating scale (NRS) ranging from no anxiety (0) to severe anxiety (10).
Time Frame: At baseline, and at 1 hour after initiation of nitrous oxide
Population: Data are included for all participants from which they were collected.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nitrous Oxide
Number analyzed (Participants) | 15
units on a scale
  Baseline | 2.50 (3.54)
  1 hour after initiation of nitrous oxide: number analyzed (Participants) | 10
  1 hour after initiation of nitrous oxide | 2.00 (3.35)
Statistical Analysis 1: Comparison: Nitrous Oxide; Test type: Other; p = 0.73, t-test, 2 sided

3. Other Pre Specified Outcome: Nausea
Description: Participant reported nausea score, using a numerical rating scale (NRS) ranging from no nausea (0) to severe nausea (10).
Time Frame: At baseline, and at 1 hour after initiation of nitrous oxide
Population: Data are included for all participants from which they were collected.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nitrous Oxide
Number analyzed (Participants) | 16
units on a scale
  Baseline | 0.25 (0.58)
  1 hour after initiation of nitrous oxide | 0.46 (1.03)
Statistical Analysis 1: Comparison: Nitrous Oxide; Test type: Other; p = 0.56, t-test, 2 sided

4. Other Pre Specified Outcome: Emesis
Description: Participant reported emesis (yes or no).
Time Frame: During administration of nitrous oxide
Population: Data are included for all participants from which they were collected.
Measure: Number; unit: participants experiencing emesis
Arm/Group | Nitrous Oxide
Number analyzed (Participants) | 16
participants experiencing emesis | 1

5. Other Pre Specified Outcome: Participant Satisfaction
Description: Participant reported score of satisfaction with nitrous oxide for labor analgesia, using a numerical rating scale (NRS) ranging from completely dissatisfied (0) to completely satisfied (100).
Time Frame: 24 hours after delivery
Population: Data are included for all participants from which they were collected.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Nitrous Oxide
Number analyzed (Participants) | 3
units on a scale | 90 [85 to 100]

6. Other Pre Specified Outcome: Crossover To Epidural
Description: Participants crossing over from nitrous oxide to epidural.
Time Frame: Initiation of nitrous oxide to completion of delivery.
Population: Data are included for all participants from which they were collected.
Measure: Number; unit: participants
Arm/Group | Nitrous Oxide
Number analyzed (Participants) | 15
participants | 8

ADVERSE EVENTS:
Arm/Group | Nitrous Oxide
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 16/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nitrous Oxide (N=16)
Pain (General disorders) | 16
Anxiety (Psychiatric disorders) | 7
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Sinus Bradycardia (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 3
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
The study was limited by its small size. Additionally, because all participants were recruited from Family Medicine clinics in Pittsburgh, these results may not be generalizable to other populations of pregnant women.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes